CLINICAL TRIAL: NCT03447405
Title: Dino Egg Mother's Voice Exposure and Speech Sound Processing in Neonatal Intensive Care Unit Infants
Brief Title: Dino Egg in Neonatal Intensive Care Unit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant not funded
Sponsor: Jonathan Slaughter (Other)
Responsible Party: Sponsor-Investigator, Jonathan Slaughter, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB18-00012
Record Dates: First submitted 2018-01-23; First posted 2018-02-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Premature Birth
Keywords: Music Therapy; NICU; Infants; multisensory processing
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Test the usability of the device (safety for the NICU was confirmed), not the effectiveness of the parents' voice delivery for the infant. Parent and nursing questionnaires about the importance of the device availability and its usability will be collected from parents and RN staff that choose to provide the feedback.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dino Egg Safety and useability (Experimental): Test the usability of the device (safety for the NICU was confirmed), not the effectiveness of the parents' voice delivery for the infant. Parent and nursing questionnaires about the importance of the device availability and its usability will be collected from parents and RN staff that choose to provide the feedback.
  Interventions: Device: Dino Egg
- Standard of Care (No Intervention)

INTERVENTIONS:
Device: Dino Egg — DINO EGG speakers, a NICU-safe and developmentally appropriate music player that delivers parent's voice to the bedside of NICU infants. The device passed NCH NICU-safe products committee and has been used in the clinical setting delivering clinical music therapy services (available at bedside to play parents' voice).
  Arms: Dino Egg Safety and useability

SUMMARY:
Dino EGG mother's voice exposure and multisensory processing in Neonatal Intensive Care Unit infants.

This is a 2 phase prospective comparative effectiveness trial of our parents' voice intervention with 290 hospitalized preterm infants.

As a part of a previous project, an early technology development award from the Nationwide Children's Hospital (NCH) Technology Office allowed us to develop 10 functioning prototypes of the DINO EGG speakers, a NICU-safe and developmentally appropriate music player that delivers parent's voice to the bedside of NICU infants. The device passed NCH NICU-safe products committee and has been used in the clinical setting delivering clinical music therapy services (available at bedside to play parents' voice).

The first phase of the current study is to test an updated prototype version of the device that replicates a previously FDA (and NCH NICU-safe products) proved device called Pacifier Activated Lullaby (PAL), used and described in IRB15-01035, but being discontinued by the company. The discontinuation is not due to safety or health benefits concerns. Therefore, no device available on the market currently exists to accomplish NICU parents' voice delivery in a consistent and safe manner, the investigators modified a 510K-approved feeding device that is no longer available and whose intellectual property rights have expired. The device's air displacement sensor, which fits into a standard NICU pacifier, allowed the investigators to deliver processed and developmentally appropriate recordings of parent's voice, contingent upon the infant producing effort to receive it. Intellectual property rights were filed for the modifications and use process through the technology transfer and legal office at NCH.

Therefore, phase I will test the usability of the device (safety for the NICU was confirmed), not the effectiveness of the parents' voice delivery for the infant. Parent and nursing questionnaires about the importance of the device availability and its usability will be collected from parents and Registered Nurse (RN) staff that choose to provide the feedback.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be Post Menstrual Age (PMA) 32 0/7-34 6/7.

Exclusion Criteria:

* Ventilation using an endotracheal tube
* Major congenital malformations
* Family history of genetic hearing loss
* Use of sedatives or seizure medications
* Presence of severe neural injury on neuroimaging (intraventricular hemorrhage grade II or IV, periventricular leukomalacia, cerebellar hemorrhage, ischemic or thrombotic injury)
* Presence of systemic inflammatory conditions (history of necrotizing enterocolitis Bell's stage IIA or above or culture-documented sepsis or meningitis).

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Usability of the device through questionaires | Through end of study completion, an average of 1 year
  We will confirm a larger scale that for preterm infants, standardized exposure to mother's voice with a contingent stimulus of non-nutritive sucking can improve the development of speech sound discrimination in the NICU. Phase I will test the usability of the device (safety for the NICU was confirmed), not the effectiveness of the parents' voice delivery for the infant. Parent and nursing questionnaires about the importance of the device availability and its usability will be collected from parents and RN staff that choose to provide the feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie L Maitre, MD,PHD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States